CLINICAL TRIAL: NCT04768504
Title: An Open-label Study of Tofacitinib for the Treatment of Refractory Immune-related Colitis from ChecKpoint Inhibitor Therapy (TRICK)
Brief Title: Tofacitinib for the Treatment of Refractory Immune-related Colitis from Checkpoint Inhibitor Therapy- TRICK Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision, due to low recruitment rate
Sponsor: Khashayar Esfahani (Other)
Responsible Party: Sponsor-Investigator, Khashayar Esfahani, Dr., Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR2108KE
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Immune-Mediated Colitis
Keywords: Immune-related adverse events; Immune-related colitis
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Tofacitinib 10 mg PO BID for 30 days
  Interventions: Drug: Tofacitinib 10 mg

INTERVENTIONS:
Drug: Tofacitinib 10 mg — Tofacitinib 10 mg PO BID for 30 days

SUMMARY:
This is a single-arm pilot study evaluating the efficacy and safety of tofacitinib in cancer patients with immune-related colitis from immune checkpoint inhibitor (ICI) therapy.

DETAILED DESCRIPTION:
Primary objective and endpoint

• Efficacy of tofacitinib in inducing clinical remission of immune related colitis, as measured by the proportion of patients who experience diarrhea resolution to grade ≤1 as per Common Terminology Criteria for Adverse Events [CTCAE] v5.0) without the requirement for additional immunosuppression (e.g., corticosteroids, biologics, or other immunosuppressors targeted for colitis) 8 weeks post-first dose of tofacitinib.

Secondary objectives and endpoints:

* Safety of tofacitinib in cancer patients with immune-related colitis, as defined by the occurrence of adverse events grade ≥3.
* Efficacy of tofacitinib in cancer patients with immune colitis as defined by endoscopic remission of colitis (a total Mayo score of ≤2) at 8 weeks.
* Efficacy of tofacitinib to induce a clinical remission of immune-related colitis as measured by the time, in days, necessary to achieve a diarrhea of grade ≤ 1 (as per CTCAE v 5.0).
* Number of patients with tumor progression at 8 weeks per iRECIST and RECIST 1.1 criteria compared to baseline scans.

Exploratory objective

• The study will collect blood samples from participants seeking to characterize the inflammatory landscape of ICI-mediated colitis and biomarkers predictive of response to tofacitinib.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Able to provide informed consent.
3. Diagnosis of a solid tumor treated with an immune checkpoint inhibitor (ICI), with the exception of colorectal cancer.
4. Exposure to an ICI (CTLA-4, PD-1, PDL-1) as part of a cancer treatment regimen within 6 months of the onset of colitis symptoms. The ICI may be used as a single agent, or in combination with other ICIs, or with chemotherapy.
5. Current diagnosis of immune-related colitis characterized by grade ≥ 2 diarrhea as per CTCAE v5.0.
6. Patients should have failed corticosteroids (at least 1mg/kg equivalent of prednisone for a minimum of 72 hours), and at least one dose of a biologic agent (i.e. either a TNFα inhibitor or an anti-integrin). Failure is defined as having ongoing grade ≥ 2 diarrhea per CTCAE v5.0.
7. Adequate hematological function, defined by:

   1. hemoglobin ≥ 90 g/L
   2. absolute neutrophil count ≥ 1.0 x 109/L
   3. lymphocyte count ≥ 0.5 x 109/L
   4. platelets ≥ 75 x 109/L
   5. PT, PTT, INR ≤ 1.5 x upper limit of normal (ULN).
8. Adequate liver function, as assessed by the Child Pugh classification score (appendix 1). Patients with scores A and B are eligible for enrollment. Patients with severe hepatic impairment (Child Pugh C) are excluded from the study.
9. Adequate renal function as defined by an estimated clearance ≥ 40 mL/min, calculated per the Cockroft-Gault formula (appendix 2).
10. Women of childbearing potential (WOCBP) are eligible if they agree to use adequate contraception while on study. If in line with the patient's preference and usual lifestyle, complete abstinence from heterosexual intercourse is acceptable. WOCBP must otherwise agree to correctly and consistently use at least one "highly effective" in addition to one "effective" contraceptive methods:

Highly effective means of contraception include the following:

* Hormonal methods of contraception including combined oral contraceptives, vaginal ring, injectables, patch, implants, and intrauterine systems (IUSs).
* Nonhormonal intrauterine devices (IUDs).
* Tubal ligation
* Vasectomy of the sole partner of a female subject
* Male condoms with spermicide

Effective means of contraception include the following:

* Diaphragm with spermicide
* Cervical cap with spermicide
* Vaginal contraceptive sponge
* Male condom without spermicide
* Female condom (a male and female condom must not be used together)

Exclusion criteria:

1. Diagnosis of a thromboembolic event (deep vein thrombosis, pulmonary embolism, embolic stroke, myocardial infarction, or peripheral arterial insufficiency) within 3 months of enrollment.
2. Diagnosis of concomitant infectious colitis (e.g. C. difficile or other bacterial source), unless the patient has finished an appropriate length of treatment with antibiotics as indicated for each diagnosis at the time of enrollment.
3. Any other grade ≥ 3 infection at the time of enrollment.
4. Prior therapy with a JAK inhibitor within 3 months preceding enrollment.
5. Use of strong inducers of CYP3A4 within 7 days of starting treatment with tofacitinib (see appendix 3).
6. Known allergy or hypersensitivity to tofacitinib, its excipients or any of the drugs used in this study (valacyclovir, heparin, trimethoprim and sulfonamides).
7. Active pregnancy or breastfeeding.
8. Patients on intravenous biologic agents for other baseline autoimmune conditions.
9. Patients having other concomitant uncontrolled irAEs at the time of enrollment which would require systemic corticosteroids or biologic immunomodulatory agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Clinical Remission of Diarrhea | 8 weeks from first dose
  Resolution of diarrhea to grade 1 or less per Common Terminology Criteria for Adverse Events

SECONDARY OUTCOMES:
Safety of tofacitinib | from first dose to 30 days post last dose
  Defined as the occurrence of Grade 3 or higher adverse events
Endoscopic remission | At 8 weeks
  per Mayo score of less or equal than 2
Time to clinical remission | from baseline to 8 weeks post first dose
  time in days to resolution of diarrhea to grade 1 or less
Tumor response status | 8 weeks from first dose
  number of patient with PD by RECIST/iRECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Khashayar Esfahani, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Sir Mortimer B Davis Jewish General Hospital - CIUSSS Centre-Ouest, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esfahani K, Hudson M, Batist G. Tofacitinib for Refractory Immune-Related Colitis from PD-1 Therapy. N Engl J Med. 2020 Jun 11;382(24):2374-2375. doi: 10.1056/NEJMc2002527. No abstract available. PMID 32521140